CLINICAL TRIAL: NCT01881867
Title: Phase 2 Study of Recombinant Glycosylated Human Interleukin-7 (CYT107) After Completion of Standard Therapy With Sipuleucel-T (Provenge®) in Pts w/ Asymptomatic or Minimally Symptomatic Metastatic Castration-Resistant Prostate Cancer(mCRPC)
Brief Title: CYT107 After Vaccine Treatment (Provenge®) in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Cancer Immunotherapy Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mac Cheever, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CITN12-03; NCI-2013-00998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN12-03 (Other: CITN); CITN12-03 IL7 (Other: Fred Hutchinson Cancer Research Center); CITN12-03 (Other: Cancer Immunotherapy Trials Network); P30CA015704 (NIH); P50CA097186 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (no therapy) (No Intervention): Patients receive no treatment (observation) after completion of standard sipuleucel-T therapy.
- Cohort II (glycosylated recombinant human interleukin-7) (Experimental): Patients receive glycosylated recombinant human interleukin-7 SC every week for 4 weeks (on days 0, 7, 14, and 21) beginning 3-7 days after completion of standard sipuleucel-T therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Glycosylated Recombinant Human Interleukin-7; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Glycosylated Recombinant Human Interleukin-7 — Given SC
  Other Names: CYT107; Glycosylated rhIL-7
  Arms: Cohort II (glycosylated recombinant human interleukin-7)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Cohort II (glycosylated recombinant human interleukin-7)

SUMMARY:
This randomized phase II trial studies how well glycosylated recombinant human interleukin-7 (CYT107) after vaccine therapy works in treating patients with castration-resistant prostate cancer that has spread to other areas of the body or has not responded to at least one type of treatment. Biological therapies, such as glycosylated recombinant human interleukin-7, may stimulate the immune system in different ways and stop tumor cells from growing. Vaccines made from white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells. It is not yet known whether glycosylated recombinant human interleukin-7 works better with or without vaccine therapy in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether CYT107 administration increases the vaccine-induced antigen-specific T-cell immune response to the sipuleucel-T fusion protein vaccine construct prostatic acid phosphatase granulocyte-macrophage colony-stimulating factor (PAP-GM-CSF) (PA2024).

SECONDARY OBJECTIVES:

I. To determine whether CYT107 administration increases the vaccine-induced antigen-specific T-cell immune response to PAP.

II. To assess the character of the T-cell immune response to PAP and PA2024. III. To determine whether CYT107 administration increases the vaccine-induced antigen-specific antibody immune responses to PAP and PA2024.

IV. To quantify the effects of CYT107 on T-cell repertoire diversity. V. To assess the effects of CYT107 on the immune competence of patients with advanced prostate cancer.

VI. To assess the clinical efficacy and tolerability of sipuleucel-T plus CYT107 compared with sipuleucel-T alone.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Patients receive no treatment (observation) after completion of standard sipuleucel-T therapy.

COHORT II: Patients receive glycosylated recombinant human interleukin-7 subcutaneously (SC) every week for 4 weeks (on days 0, 7, 14, and 21) beginning 3-7 days after completion of standard sipuleucel-T therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 53 weeks. Patients are followed by phone, once a year, after completion of Week 53 for overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic or minimally symptomatic metastatic castration-resistant prostate cancer (mCRPC)
* Patients must have successfully completed therapy with sipuleucel-T within 3-7 days of planned CYT107 study drug treatment
* Assessable disease with a positive bone scan and/or measurable disease on computed tomography (CT) scan and/or magnetic resonance imaging (MRI) of the abdomen and pelvis
* Prior orchiectomy or must be on ongoing luteinizing hormone-releasing hormone (LHRH) agonist or antagonist (e.g., degarelix) therapy
* No ongoing anti-androgen therapy; patients must be off anti-androgen therapy for at least 30 days
* Patients receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease prostate specific antigen (PSA) levels (e.g. saw palmetto, PC-SPES), or any systemic corticosteroid, must discontinue the agent for at least 30 days prior to study treatment
* Absolute neutrophil count (ANC) >= 1500/uL
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Hemoglobin >= 10 g/dL
* Platelets >= 100,000/mcL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance >= 60 mL/min by the Cockcroft-Gault equation
* Testosterone =< 50 ng/dL (documented at any time while on LHRH agonist or antagonists or s/p orchiectomy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 or a Karnofsky performance status of >= 80%
* Life expectancy of at least 6 months
* Prior local radiation therapy must be completed at least 30 days prior to enrollment and the patient must have recovered from all toxicity
* Prior "systemic" radiopharmaceuticals (strontium, samarium, radium 223 dichloride) must be completed >= 8 weeks prior to enrollment
* Patients must agree to use 2 methods of adequate contraception for the duration of study participation, and for four months after discontinuing therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior chemotherapy for castration resistant prostate cancer; neoadjuvant chemotherapy and chemotherapy given for hormone sensitive prostate cancer are allowed
* Prior investigational immunotherapy
* Prostate cancer pain requiring regularly scheduled narcotics
* Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression
* Current treatment with systemic steroid therapy (inhaled/topical steroids are acceptable); systemic corticosteroids must be discontinued for at least 30 days prior to first CYT107 injection
* Known central nervous system metastases
* Documented cirrhosis or documented acute hepatitis; Note: a positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb] positive and hepatitis B core antibody [HBcAb] negative), or a fully resolved acute hepatitis B virus (HBV) infection is not an exclusion criterion
* History of severe asthma, as defined by prior or current use of systemic corticosteroids for disease control, with the exception of physiological replacement doses of cortisone acetate or equivalent, as defined by a dose of 10 mg or less
* Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves
* Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months)
* Concurrent or prior malignancy except for the following:

  * Adequately treated basal or squamous cell skin cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* Known human immunodeficiency virus (HIV) or other history of immunodeficiency disorder; HIV-positive patients on combination antiretroviral therapy are ineligible
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g. infectious) illness
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of CYT107 hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CYT107
* Patients who have received prior immunosuppressive therapy within 30 days prior to enrollment
* Active (as defined by requiring immunosuppressive therapy) or history of clinically significant autoimmune disease (as defined by previously requiring immunosuppressive therapy)
* Patients who have received hepatotoxic drugs less than 7 days prior to enrollment
* Patients who have received prior biologic agents less than 30 days prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have a history of any hematopoietic malignancy
* History of pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD), (forced expiratory volume [FEV] > 60% of predicted for height and age required in patients with prolonged smoking history or symptoms of respiratory dysfunction)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, Principal Investigator — Cancer Immunotherapy Trials Network; Martin A. Cheever, Study Director — Fred Hutchinson Cancer Research Center/Cancer Immunotherapy Trials Network
Locations (16):
- United States (16):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I (no Therapy): Patients receive no treatment (observation) after completion of standard sipuleucel-T therapy through week 53.
- Cohort II (Glycosylated Recombinant Human Interleukin-7): Patients receive glycosylated recombinant human interleukin-7 SC every week for 4 weeks (on days 0, 7, 14, and 21) beginning 3-7 days after completion of standard sipuleucel-T therapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed post-active 4 week treatment for duration of study, 53 weeks.
  Glycosylated Recombinant Human Interleukin-7: Given SC
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Started | 26 | 28
Completed | 14 | 15
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7) | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (7.6) | 67.6 (7.9) | 66.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Quantification of T-cell Responses to Prostatic Acid Phosphatase Granulocyte-macrophage Colony-stimulating Factor (PAP-GM-CSF), Assessed by Quantification of Interferon Gamma Levels Measured Using Enzyme-linked Immunospot (ELISPOT)
Description: The Mann-Whitney-Wilcoxon (MWW) test will be used as part of the statistical analysis to determine quantification of T-cell responses to prostatic acid phosphatase granulocyte-macrophage colony-stimulating factor (PAP-GM-CSF), as assessed by quantification of interferon gamma levels measured using enzyme-linked immunospot (ELISPOT). The power is roughly equivalent to that based on the t-test.
Time Frame: Day 70 (week 11)
Measure: Mean (Standard Deviation); unit: T cell spots per 300,000 PBMC
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 15 | 25
T cell spots per 300,000 PBMC | 212.2 (111.97) | 199.68 (182.4)

2. Secondary Outcome: Change in Bystander Antigen Specific Immune Responses, Measured by Interferon Gamma Production in Response to Various Antigens as Quantified by Enzyme-linked Immunospot (ELISPOT)
Description: Bystander antigen specific immune responses will be assessed to other ongoing and nascent antitumor responses (e.g., preferentially expressed antigen in melanoma, cancer/testis antigen 1B and/or tumor protein p53), additional tumor antigens specific to prostate cancer (e.g., prostate specific antigen [PSA] and/or prostate-specific membrane antigen), and memory viral responses (influenza A and cytomegalovirus, Epstein-Barr virus and influenza virus-derived peptides) using the interferon gamma ELISPOT assay.
Time Frame: Baseline to up to week 53
Population: No subjects were tested for bystander antigen specific immune responses because there was no indication that there was an enhanced response in the primary objective.
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Circulating Tumor Cells
Description: Enumerated by the approved Veridex assay.
Time Frame: Baseline to up to week 53
Population: Cohort 1: 16 subjects analyzed at Week 01 and 8 subjects analyzed at Week 53. Cohort 2: 22 subjects analyzed at Week 01 and 5 subjects analyzed at Week 53.
Measure: Mean (Standard Deviation); unit: Circulating Tumor Cells
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 16 | 22
Circulating Tumor Cells
  Week 01 | 2.56 (7.88) | 1.45 (2.97)
  Week 53: number analyzed (Participants) | 8 | 5
  Week 53 | 2.63 (5.97) | 0 (0)

4. Secondary Outcome: Change in Number of Peripheral Blood Mononuclear Cell (PBMC) Subsets and T Lymphocyte Subsets
Description: The absolute fold change from baseline of CD3+ cells
Time Frame: Week 11
Population: Subjects for whom whole blood was collected at protocol specified timepoints
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 14 | 22
fold change
  Week 06: number analyzed (Participants) | 14 | 21
  Week 06 | 1.05 (0.29) | 2.33 (1.02)
  Week 11: number analyzed (Participants) | 9 | 22
  Week 11 | 1.21 (0.34) | 1.77 (0.55)

5. Secondary Outcome: Change in Prostate Specific Antigen (PSA) Kinetics.
Description: The change in prostate specific antigen (PSA) kinetics will be evaluated according to the recommendations from PSA Working Group (PSAWG). Analysis of PSA doubling time
Time Frame: Baseline to up to week 53
Population: Study participants who provided blood for PSA testing and analysis
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 24 | 28
Weeks | 46.82 [17.49 to 76.15] | 8.15 [-18.79 to 35.09]

6. Secondary Outcome: Change in Vaccine-induced Antigen-specific Antibody Immune Response to Prostatic Acid Phosphatase (PAP)
Description: Will be measured by change in immunoglobulin G (IgG) and immunoglobulin M (IgM) levels quantified by standard enzyme-linked immunosorbent assay (ELISA). Fold change from baseline in week 6 titer
Time Frame: Baseline to up to week 6
Population: Participants who provided blood samples to test for antibody levels to PAP
Measure: Median (Full Range); unit: fold change
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 24 | 28
fold change
  IgG-IgM levels | 8 [0.5 to 256] | 8 [1 to 64]
  IgG levels | 4 [1 to 32] | 2 [1 to 128]

7. Secondary Outcome: Overall Survival
Description: Number of participants that have survived
Time Frame: Up to 5 years
Measure: Number; unit: Participants
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
Number analyzed (Participants) | 26 | 28
Participants | 22 | 25

ADVERSE EVENTS:
Time Frame: 53 weeks
Arm/Group | Cohort I (no Therapy) | Cohort II (Glycosylated Recombinant Human Interleukin-7)
All-Cause Mortality (participants affected / at risk) | 4/26 | 3/28
Serious Adverse Events (participants affected / at risk) | 2/26 | 8/28
Other Adverse Events (participants affected / at risk) | 26/26 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (no Therapy) (N=26) | Cohort II (Glycosylated Recombinant Human Interleukin-7) (N=28)
Acute Kidney Injury (Investigations) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 1 (1)
Acute kidney injury (Investigations) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypernatremia (Investigations) | 0 (0) | 1 (1)
Hypokalemia (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (no Therapy) (N=26) | Cohort II (Glycosylated Recombinant Human Interleukin-7) (N=28)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left forearm hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (Blood and lymphatic system disorders) | 5 (5) | 7 (8)
neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
General weakness (General disorders) | 1 (1) | 0 (0)
Worsening of osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Site injection reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalized pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
lower extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
scrotal edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
hyponatremia (Investigations) | 4 (4) | 0 (0)
Bilateral pedal edema (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 2 (2) | 4 (4)
hyperglycemia (Endocrine disorders) | 2 (2) | 1 (1)
anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Decreased absolute neutrophil count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 2 (2)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
right groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gut disturbance (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hand spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Left ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left hip pain/leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Pain (Nervous system disorders) | 1 (1) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (41)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (3)
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (15)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
MRSA UTI (Infections and infestations) | 0 (0) | 1 (1)
Decreased platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Elevated ALT (Investigations) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
achy joints (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Elevated AST (Investigations) | 0 (0) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Lower extremity edema (Vascular disorders) | 0 (0) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Great toe injury with bleeding beneath nail (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased lymphocytes (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Fever (Immune system disorders) | 0 (0) | 1 (1)
Flu-like symptoms (Immune system disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gynecomastia (Endocrine disorders) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 0 (0) | 1 (1)
Hot flashes (Endocrine disorders) | 0 (0) | 1 (1)
Hypophosphotemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated creatinine (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
chills (Immune system disorders) | 0 (0) | 1 (1)
Right-side mid-back pain with degenerative changes (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain with swelling due to enlarged cervical lymph nodes (Endocrine disorders) | 0 (0) | 1 (1)
Head cold (Infections and infestations) | 0 (0) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Difficulty sleeping due to discomfort from great toe injury (Nervous system disorders) | 0 (0) | 1 (1)
Neck pain with degenerative changes (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Hyperesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Right sciatic discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Pain right scapula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Presyncopal episode (General disorders) | 0 (0) | 1 (1)
itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritic rash over right shin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritic rash over buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema left arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fainting episode (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT01881867/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT01881867/SAP_001.pdf